CLINICAL TRIAL: NCT05232058
Title: FRENCH OBSERVATORY OF ACUTE HEART FAILURE-2
Acronym: OFICA2
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A03222-55
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2009, OFICA 1 provided a snapshot of the management of acute heart failure in France.

Over the past 10 years, practitioners have observed a change in the profiles of hospitalized patients and it is necessary to specify the evolution of these characteristics, especially since the recommendations concerning management have changed significantly; this is the objective of this observatory.

Like patients suffering from chronic diseases such as diabetes or asthma, heart failure patients are therefore at the center of their management. Compliance is improved when patients have understood the reason for the prescription. Ideally, compliance should not be achieved by respecting externally imposed norms, but rather by respecting norms that are understood, adapted, personalized and accepted.

A self-questionnaire will thus be given to patients on the day of inclusion in the study.

In heart failure patients with an average age of 80 years, systematic screening for cognitive disorders using a simple test recommended by the French National Authority for Health (Haute Autorité de Santé), the codex test, will make it possible to offer more appropriate care if necessary (geriatric or neurology consultation).

Finally, follow-up at 3 months and at 1 and 2 years will be carried out by matching with data from the National Health Data System (SNDS)

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized, regardless of the initial mode of admission, with acute heart failure (de novo heart failure or decompensation of chronic heart failure) of any severity and corresponding to one of the following clinical situations :

  1. Pulmonary edema, hypertensive or not
  2. Congestive heart failure (pulmonary congestion, peripheral oedema)
  3. Cardiogenic shock
  4. High output heart failure
  5. Isolated right heart failure
* Patient who agreed to participate in the study

Exclusion Criteria:

* Expressed refusal to participate in the study
* Scheduled hospitalization for assessment
* Surgical context (immediate postoperative period)
* Diagnosis of acute heart failure reversed to another diagnosis before end of hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only inpatient facilities with at least one cardiology unit will be selected. The inclusion services will be restricted within these institutions to cardiology services, intensive care units, door beds, and internal medicine and geriatric servicesThe diagnosis of acute heart failure will be made by the investigating physician in each center, according to the clinical and paraclinical elements at his disposal.
Sampling Method: Non-Probability Sample
Enrollment: 1593 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Analyze survival during hospitalization | Trough length of hospitalization, an average of 10 days
  Rate of death during hospitalizaton

SECONDARY OUTCOMES:
Analyze survival at 2 years after hospitalisation | 2 years after hospitalisation
  Rate of death at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lariboisière, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No